CLINICAL TRIAL: NCT02383134
Title: The Maximum Effective Needle-to-Nerve Distance for Anesthetic Ultrasound-Guided Supraclavicular Brachial Plexus Block
Brief Title: Maximal Distance for Successful Supraclavicular Block
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tunisian Military Hospital (Other)
Responsible Party: Principal Investigator, Dr trabelsi walid, associate professor, MD, Tunisian Military Hospital
Other Study IDs: TunisianMH
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-03

CONDITIONS: Regional Anesthesia; Ultrasound; Supraclavicular Block

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The achievement of peripheral nerve block requires several needle passes, with each of them being at risk of causing nerve injury either by direct trauma or intraneural injection even with the use of the ultrasound.

The ultrasound guided supraclavicular brachial plexus block is known to be at risk of pneumothorax and / or nerve injury.

This study is designed to determine the maximal effective distance away from the nerve for the injection to be effective.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* 18-85 years of age, inclusive
* surgery less than 3 hours

Exclusion Criteria:

* contraindications to brachial plexus block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the area)
* existing neurological deficit in the area to be blocked
* pregnancy
* history of neck surgery or radiotherapy
* inability to understand the informed consent and demands of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing upper limb surgery surgery (hand, forearm, elbow)
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Success of the ultrasound guided supraclavicular block at 30 minutes after injection at a specific distance of the needle tip from the outer sheeth of the nerve | 30 minutes

SECONDARY OUTCOMES:
•The onset time of sensory and motor block | the block success will be assessed for each patient every 5 min for 30 mins in the operating room beginning when the needle exits the skin
The proportion of inadequate and failed blocks. | the block success will be assessed for each patient every 5 min for 30 mins in the operating room beginning when the needle exits the skin
The presence of other complications such as hematoma, infection, pneumothorax. | up to 48 hours post operative.